CLINICAL TRIAL: NCT05145127
Title: AN OPEN-LABEL EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY, TOLERABILITY, AND EFFICACY OF MARSTACIMAB PROPHYLAXIS IN SEVERE (COAGULATION FACTOR ACTIVITY <1%) HEMOPHILIA A PARTICIPANTS WITH OR WITHOUT INHIBITORS OR MODERATELY SEVERE TO SEVERE HEMOPHILIA B PARTICIPANTS (COAGULATION FACTOR ACTIVITY ≤2%) WITH OR WITHOUT INHIBITORS
Brief Title: Open-Label Extension Study of Marstacimab in Hemophilia Participants With or Without Inhibitors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7841007; PHASE 3 ANTI-TFPI OLE (Other: Alias Study Number); 2022-500470-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Factor VIII Inhibitor; Factor IX Inhibitor; PF-06741086; Marstacimab; Anti-TFPI
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06741086 (Experimental): For participants aged ≥12 years 300 milligrams(mg) subcutaneous (sc) loading dose followed by 150 mg sq once weekly (qw). 300 mg sc qw is prescribed for participants who meet dose escalation criteria.
  For participants aged ≥6 to <12 years is marstacimab 150 mg SC for initial loading dose followed by 75 mg SC QW. 150 mg sc qw is prescribed for participants who meet dose escalation criteria.
  Interventions: Drug: PF-06741086

INTERVENTIONS:
Drug: PF-06741086 — For participants aged ≥12 years 300 milligrams(mg) subcutaneous (sc) loading dose followed by 150 mg sq once weekly (qw). 300 mg sc qw is prescribed for participants who meet dose escalation criteria.
  For participants aged ≥6 to <12 years is marstacimab 150 mg SC for initial loading dose followed by 75 mg SC QW. 150 mg sc qw is prescribed for participants who meet dose escalation criteria.
  Other Names: marstacimab

SUMMARY:
Study B7841007 is an open-label extension study to assess the long-term safety, tolerability, and efficacy of prophylaxis treatment with marstacimab in participants who did not require "Early Termination" from the Phase 3 Study B7841005 and from the Phase 3 Study B7841008.

Study B7841005: approximately 145 adolescent and adult participants 12 to <75 years of age with severe hemophilia A or moderately severe to severe hemophilia B (defined as FVIII activity <1% or FIX activity ≤2%, respectively) with or without inhibitors are expected to be enrolled in Study B7841005 during which they will receive prophylaxis (defined as treatment by SC injection of marstacimab).

Study B7841008: this is an ongoing Phase 3, open-label study in pediatric participants <18 years of age with severe hemophilia A (FVIII Coagulation Factor Activity <1%) or moderately severe to severe hemophilia B (FIX Coagulation Factor Activity ≤2%). A sequential approach will be used in enrolling at least 100 pediatric participants, at least 20 of which will be aged ≥12 to <18 years and at least 80 participants will be aged ≥1 to <12 years. At the start of study B7841008, the dosing and data available in adolescent and adult participants in Study B7841005 supported the initiation of B7841008 study in participants aged ≥12 to <18 years. Subsequently, additional safety and efficacy data from adolescent participants in Study B7841005 became available for benefit/risk assessment in support of dosing participants aged ≥6 to <12 years. Based on the positive benefit/risk assessment conducted by both internal Pfizer review and eDMC review, dosing of the ≥6 to <12 years age group was initiated in June 2023 in B7841008 Study. Data from participants ≥6 years from B7841008 Study and Study B7841005 will support the dosing of participants aged ≥1 to <6 years.

All participants will be provided the prefilled pen (PFP) for administration of marstacimab in the study. Use of the prefilled syringe (PFS) will be permitted at the investigator's discretion for those participants who have difficulty with administration of the PFP. Additionally, participants will be provided the PFS for use in this study in countries where the PFS is anticipated to be the only presentation available commercially. An optional, open-label, single arm, substudy using the PFP was completed in the first 23 participants rolled over from Study B7841005 who agreed to participate in the substudy.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have a minimum body weight as defined by parent studies
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Participants have successfully completed participation in parent studies, defined as did not require "Early Termination"

Exclusion Criteria:

* Previous or current treatment for or history of coronary artery disease, venous or arterial thrombosis (CTCAE Grade >3), or ischemic disease (except catheter-associated thrombosis)
* Abnormal renal function as defined by eGFR <30 mL.min/1.73 m(2)
* Known planned surgical procedure during the planned study period
* Unstable hepatic function as determined by the Investigator clinical assessment and review of the participant's most recent laboratory results, which would make the participant inappropriate for the study
* For participants known to be HIV+, worsening disease status as determined by the Investigator clinical assessment and review of participant's most recent laboratory results, to include recent locally available CD4 count (if available), which would make the participant inappropriate for the study
* Regular, concomitant therapy with immunomodulatory drugs (eg, IVIG, and routine systemic corticosteroids, rituximab)
* Ongoing or planned use of immune tolerance induction or prophylaxis with FVIII or FIX replacement during the study
* Participation in other study involving investigational drug(s) or investigational vaccine(s) within 30 days or 5 half-lives prior to or during study participation, with the exception of participation in parent studies
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the Investigator, and their respective family members

Ages: 1 Year to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants only
Enrollment: 245 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of subject reporting Adverse Events | Baseline up to 7 years
Number of subjects reporting Serious Adverse Events | Baseline up to 7 years
Incidence and severity of thrombotic events | Baseline up to 7 years
Incidence and severity of thrombotic microangiopathy | Baseline up to 7 years
Number of subjects reporting Disseminated intravascular coagulalopathy/consumption coagulopathy | Baseline up to 7 years
Incidence of clinically significant persistent NAb against marstacimab | Baseline up to 7 years
Incidence and severity of injection site reaction | Baseline up to 7 years
Clinically significant changes in vital signs from baseline | Baseline up to 7 years
Incidence of clinically significant laboratory value abnormalities | Baseline up to 7 years
Incidence of severe hypersensitivity and anaphylactic reactions | Baseline up to 7 years

SECONDARY OUTCOMES:
Annualized rate of bleeding episodes | Baseline up to 7 years
  Derived for each subject for each treatment period by using the following formula: ABR = number of bleeds requiring treatments/ (days on treatment period / 365.25)
Total coagulation factor product consumption | Baseline up to 7 years
Incidence of joint bleeds | Baseline up to 7 years
Incidence of spontaneous bleeds | Baseline up to 7 years
Incidence of target joint bleeds | Baseline up to 7 years
Incidence of total bleeds (treated and untreated) | Baseline up to 7 year
Change in joints measured by the HJHS | Baseline up to 7 years
  Change in joints as measured by the HJHS for participants ≥4 years of age
Change in number of target joints per subject from baseline | Baseline up to 7 years
Changes in Health Utilities Measure questionnaire data | Baseline up to 7 years
Changes in Haem-A-QoL questionnaire data for participants ≥17 years of age | Baseline up to 7 years
Changes in Haemo-QoL questionnaire data | Baseline up to 7 years
  Haemo-QoL CII (Ages 8 to <12 years), Haemo-QoL (Ages 12 to <17),
Total bypass product consumption | Baseline up to 7 years
Changes in EQ-5D questionnaire data | Baseline up to 7 years
  EQ-5D-Y Proxy (Ages ≥ 4 to ≤ 6 years), EQ-5D-Y Self (Ages ≥ 7 to ≤ 11 years), EQ-5D-5L (Ages ≥12)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Northwell Health HTC, New Hyde Park, New York
  - Washington Institute for Coagulation d/b/a WACBD, Seattle, Washington
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
- China (6):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Hôpital Universitaire Necker Enfants Malades, Paris, France
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- India (4):
  - Nirmal Hospital Pvt Ltd., Surat, Gjuarat
  - K.J. Somaiya Hospital, Mumbai, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
- Sheba Medical Center, Ramat Gan, Central District, Israel
- Italy (2):
  - AOU Policlinico Umberto I, Roma, RM
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
- Japan (5):
  - Nagoya University Hospital - Transfusion Medicine, Nagoya, Aichi-ken
  - Nagano Children's Hospital, Azumino, Nagano
  - Nara Medical University Hospital, Kashihara, Nara
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - Hiroshima University Hospital, Hiroshima
- Mexico (2):
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatán S., Mérida, Yucatán
- Sultan Qaboos University Hospital, Muscat, Oman
- Serbia (2):
  - Institute for Mother and Child healthcare "Dr Vukan Cupic", Belgrade
  - Clinical Center Nis, Niš
- South Africa (4):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Worthwhile Clinical Trials, Benoni
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
- South Korea (4):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi[seoul]
  - Kyungpook National University Hospital, Daegu, Taegu-kwangyǒkshi
- Spain (4):
  - Hospital Universitario A Coruna, A Coruña
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (2):
  - ChangHua Christian Hospital, Changhua, Changhua County
  - Taichung Veterans General Hospital, Taichung
- Turkey (Türkiye) (8):
  - Acibadem Adana Hospital, Adana
  - Hacettepe University Faculty of Medicine, Ankara
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Gaziantep University Şahinbey Research and Practice Hospital, Gaziantep
  - Istanbul University Oncology Institute, Istanbul
  - Ege University Faculty of Medicine, Izmir
  - Erciyes University Faculty of Medicine, Kayseri
  - Ondokuz Mayıs University Healthcare Practice and Research Center, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841007